## CONSENT BY PATIENT FOR CLINICAL RESEARCH

| Version No.: 01<br>Version Date: 11th JULY 2022 |
|---|
| I, |
| hereby agree to take part in the clinical research specified below: |
| Title of Study: ACCELERATED RECOVERY FOLLOWING OPIOID-FREE ANAESTHESIA IN SUPRATENTORIAL CRANIOTOMY |
| The nature and purpose of which has been explained to me by |
| Dr(Name & Designation of Doctor) |
| and interpreted by(Name & Designation of Interpreter) to the best of his/her ability inlanguage/dialect. |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per participant information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent on my own free will to participate in the clinical research specified above. |
| I understand that I can withdraw from this clinical research at any time without assigning any reason whatsoever and in such a situation shall not be denied the benefits of usual treatment by the attending doctors. |
| Date: Signature or Thumbprint (Patient) |
| IN THE PRESENCE OF |
| Name |
| Identity Card No. Signature (Witness for Signature of Patient) |
| Designation |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research. |
| Date |

CONSENT BY PATIENT R.N.
FOR Name
CLINICAL RESEARCH Sex

Age Unit

BK-MIS-1117-E02